CLINICAL TRIAL: NCT06887153
Title: Perioperative Multimodal Analgesia Practices and Associated Acute Postoperative Pain in Patients Undergoing Major Surgery at Mulago National Referral Hospital
Brief Title: Multimodal Analgesia Utilization and Acute Postoperative Pain After Major Surgery at Mulago National Referral Hospital
Status: Recruiting | Type: Observational
Sponsor: Makerere University (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: MAK-SOMREC-2024-920
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Pain
Keywords: Perioperative; Multimodal Analgesia; Acute Postoperative Pain; Major Surgery
MeSH Terms: conditions — Pain; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to understand the approach to pain management before, during, and after surgery at Mulago National Referral Hospital. It is focussed on adult patients undergoing major surgery. The main questions it aims to answer are:

* How often are combinations of pain medications utilised before, during and after surgery?
* Do combinations of pain medications result in better pain control after surgery compared to single pain medications?

Information on pain medications will be obtained from patient records. Patients will be asked to rate their pain after surgery every 6 hours for 24 hours.

DETAILED DESCRIPTION:
Study Objectives:

Primary Objectives

* To determine the prevalence of perioperative multimodal analgesia practices among adult patients undergoing elective major surgery at Mulago National Referral Hospital.
* To determine the association between perioperative multimodal analgesia practices and acute postoperative pain among adult patients undergoing elective major surgery at Mulago National Referral Hospital.

Secondary Objective - To determine factors associated with perioperative multimodal analgesia practices at Mulago National Referral Hospital.

Study site: Mulago National Referral Hospital, the largest public hospital in Uganda with a bed capacity of 1500.

Study area: Post Anaesthesia Care Units of the Main Operating Theatre Complex and five inpatient surgical units i.e., Colorectal, Upper Gastrointestinal/Hepatobiliary, Spine, Thoracic, Orthopaedic

Study Population: All adult patients undergoing elective major surgeries in the five surgical units during the study period who meet the eligibility criteria.

Sample size assessment: calculated using the Kish Leslie (1965) formula. Adjusted for a 10% loss to follow up rate and clustering with a design effect of 1.5.

Sampling procedure: Based on monthly surgical averages, participants will be grouped as follows: Colorectal - 105 patients, Upper Gastrointestinal/Hepatobiliary - 84 patients, Spine - 112 patients, Orthopaedic - 126 patients, Thoracic - 22 patients. Consecutive sampling will be done in each of the surgical units until the desired sample size is attained.

Study procedure:

* The principal investigator or research assistants will visit the patients the evening before their scheduled surgery to screen for eligibility and obtain informed consent.
* Data on patient socio-demographics, ASA status, clinical diagnosis, type of scheduled surgery, and performance of a preoperative anaesthetic assessment will be abstracted from the patient's chart.
* Enrolled patients will be asked about any history of chronic (≥3 months) pain and use of analgesics.
* The patient will be asked about the presence of preoperative pain. If in pain, a baseline assessment will be performed using the Numeric Rating Scale, which will be physically presented to the patient. The numbers on the scale and what levels of pain they represent will be explained to the patient. The patient will then be asked to choose a number on the scale that best represents their current level of pain. Either the patient or the research assistant will circle this.
* All systemic analgesic medications (drug class, agent, dosage, frequency, route of administration, prescriber) and regional analgesic techniques (the name of the technique, cadre of the performer of the technique, and drug(s) given, including dosage and frequency) utilised in the preoperative period will be recorded.
* Upon admission to the PACU after the surgery, all systemic analgesic medications, regional analgesic techniques, and medications utilised in the intraoperative phase will be abstracted from the patient's anaesthetic chart. Additional data collected will include the cadre of the anaesthesia provider, i.e. anaesthesiologist, anaesthetic officer or anaesthesia resident and their years of practice or year of training, type of anaesthetic used, i.e. general anaesthesia, spinal anaesthesia, epidural anaesthesia or a combination of spinal and epidural anaesthesia, peripheral nerve blocks, intravenous regional anaesthesia, type of surgery performed and duration of the surgical procedure.

Postoperatively:

- All the systemic analgesic medications and regional analgesic techniques utilised in the postoperative period will be abstracted from the patient's files.

9. Pain intensity after surgery will be measured using the Numeric Rating Scale. The nurse or doctor on duty will be informed if a patient is found with an NRS of ≥4. The research assistants will follow up to ensure that interventions to relieve the patient's pain have been instituted.

Data collection and management Research assistants will undergo data collection training for three days. The abstraction form will be pre-tested before actual data collection on 10 participants who will not be part of the study. Questions will then be refined to ensure their clarity and relevance during the data collection process. All completed forms will be cross-checked for completeness by the Principal Investigator daily. Any errors, incompleteness, or incoherence will be addressed before data storage and entry.

Data will be entered into REDCap electronic data capture software with programmed data checks. The database will be stored on a password-locked hard drive, and the principal investigator's Google Drive will be used as a backup. Data cleaning will be done weekly to ensure quality data is available for analysis.

Data Analysis Data analysis will be carried out using Stata software (version 17). Univariable analysis will be achieved using frequencies with their proportions for categorical data, means with standard deviations for continuous variables with normal distribution, and medians with their interquartile ranges for continuous data with skewed distribution.

Objective 1: To determine the prevalence of perioperative multimodal analgesia practices in adult patients undergoing elective major surgery at Mulago National Referral Hospital.

Descriptive statistics will be used to describe the systemic and/or regional analgesic medications used in the perioperative period (multimodal analgesia practices). Frequencies with their proportions, means with standard deviations, and medians with their interquartile ranges will be reported appropriately. The results will be presented in tables, graphs and charts.

Objective 2 and secondary objective Binary logistic regression will be used to evaluate the association between individual independent variables (including perioperative multimodal analgesia practices) and acute postoperative pain. Variables with a p-value of less than 0.2 in the bivariable analysis will be used in the multivariable analysis. Crude odds ratio (cOR) and their 95% confidence intervals will be reported.

Multivariable logistic regression will be used to evaluate the association between perioperative multimodal analgesia practices and acute postoperative pain, adjusting for other independent variables and controlling for interaction and confounding. Adjusted odds ratios (aOR) and their 95% confidence intervals will be reported. The statistical significance in this study will be determined at a p-value less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years
* Scheduled for elective orthopaedic, abdominal and thoracic surgeries
* In the selected operating theatres during the study period

Exclusion Criteria:

* Reduced levels of consciousness or neurological deficits
* ASA >III

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who present for surgical treatment at Mulago National Referral Hospital, Kampala City, Uganda
Sampling Method: Non-Probability Sample
Enrollment: 449 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2025-06-17 (Estimated); Study Completion 2025-07-17 (Estimated)

PRIMARY OUTCOMES:
patient-reported acute postoperative pain levels | Postoperative pain will be assessed at 0, 6, 12, 18, and 24 hours postoperatively.
  This will be measured using an 11-point Numeric Rating Scale (NRS) ranging from 0 (no pain) to 10 (worst pain). Pain intensity will be graded as mild (NRS: 1-3), moderate (NRS: 4-6), and severe (NRS: 7-10).

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel S. Aporu, MBChB, Principal Investigator — Makerere University
Locations (1):
- Mulago National Referral Hospital, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 6 months after publication upto 2 years after publication
Access Criteria: Request must be reasonable. In case of intended statistical analyses, an institutionally approved proposal must be presented.